CLINICAL TRIAL: NCT01346527
Title: Maternal Lipid Metabolism and Neonatal Heart Function in Diabetes
Brief Title: Fat Metabolism in Pregnancy and Neonatal Heart Function in Diabetes
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sponsor
Other Study IDs: 10-12828
Record Dates: First submitted 2011-04-29; First posted 2011-05-03 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Type 2 Diabetes; Pregnancy
Keywords: diabetes; pregnancy; left ventricular dysfunction; neonatal; lipid; lipotoxicity; neurodevelopment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Maternal and umbilical cord serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Type 2 diabetes: 1. Women will be diagnosed with type 2 DM (pre-gestational, White classification B or C class). Since the majority of women with B or C class DM are on insulin therapy in our clinic, we will recruit only women on insulin therapy (i.e. no oral diabetes medications).
  2. HbA1C ≤ 8 for greater than 3 months32, 33.
  3. All women will have confirmed singleton pregnancies.
  4. Receive care at the Women's Health Clinic at Barnes Jewish Hospital.
  5. Pre-pregnancy BMI is anticipated to be >30 (i.e. obese) from the data regarding the patient population of our clinic. Women with pre-pregnancy BMI between 23-40 will be included.
- Healthy, obese pregnant controls: 1. No diagnosis of type 1 or 2 diabetes or previous gestational DM.
  2. Women with pre-pregnancy BMI between 30-45: control participants will be BMI matched to women with DM.
  3. A normal routine, standard of care 1 hour 50 gram gestational diabetes screen.
  4. Receive care at the Women's Health Clinic at Barnes Jewish Hospital.
  5. Patients will have a singleton pregnancy with no fetal abnormalities (as determined by routine standard of care ultrasonography).
- Healthy, Lean Controls: No diagnosis of type 1 or 2 diabetes or previous gestational DM. 2) Women with pre-pregnancy BMI between 21-25.9 3) A normal routine, standard of care 1 hour 50 gram gestational diabetes screen.

SUMMARY:
Background: The health of the next generation is likely programmed in the womb (i.e.in utero), and our understanding of how that programming happens will allow us to favorably influence the health of future generations. The focus of this proposal is to examine the effect of in utero programming on heart function in children born to women with type 2 diabetes (T2DM). Specifically, neonates born to diabetic women have abnormal heart structure and weaker heart function at birth, which may predispose them to long-term heart problems in childhood, adolescence and adulthood. At present, the reason for these heart abnormalities in children born to women with diabetes is unknown and is the focus of this proposal.

Objective(s) and Hypothesis(es): The objectives are to examine the relationships among maternal lipid (fatty acid, triglyceride, very low density lipoprotein) metabolism and neonatal heart structure and function in diabetes and to identify clinical markers during pregnancy for heart dysfunction in infants born to diabetic women. The overall hypothesis is that maternal lipid metabolism is abnormal in diabetes, and this metabolic dysregulation increases fatty acid delivery to the fetus in utero and leads to abnormal accumulation of lipid in the fetal heart, resulting in altered neonatal heart structure and function in infants born to diabetic women. In addition, the investigators hypothesize that decreased maternal fatty acid oxidation (fat "burning") rate, elevated lipolytic (fat breakdown) rate and elevated blood total free fatty acid level predicts abnormal neonatal heart structure and function in infants born to women with type 2 diabetes.

Methods and Procedures: The investigators will test these hypotheses by using clinical metabolism studies (infusion of stable isotope labeled fatty acid, serial blood and breath sampling, and mass spectrometry) to quantify whole-body fat (fatty acid oxidation, lipolysis, and serum fatty acid , triglycerides, VLDL-cholesterol levels) metabolism in 25 diabetic women during the 3rd trimester of pregnancy, and compare these lipid metabolism kinetics to 25 body mass index matched healthy non-diabetic women during pregnancy and determine if alterations in maternal lipid metabolism predict abnormal neonatal heart function in children born to these women.

Potential Impact: Type 2 diabetes is an epidemic in the United States and is steadily increasing worldwide. Diabetes has detrimental health effects in pregnant women and in their offspring. The investigators know that children born to women with diabetes have an increased risk for developing diabetes, obesity and cardiovascular disease, than children born to healthy women. This proposal will address an important knowledge gap regarding the role of maternal lipid (and potentially other nutrients) metabolism on the cardiovascular health of the global and increasing population of children born to diabetic women. Findings from this project will be novel and innovative, and will likely point to clinical interventions that target and correct lipid and other metabolic abnormalities in women with pre-gestational diabetes. The impact will be great because the long-term goal is to ameliorate heart problems in children born to diabetic (both pre-gestational and gestational) women. In addition, this project will establish a small cohort of children that can be followed long-term to address novel questions about the progression of heart and other metabolic abnormalities in children born to diabetic women.

DETAILED DESCRIPTION:
Background: In the United States, there are approximately 1.2 million children born to women with diabetes mellitus (DM) each year. This number is increasing due to the epidemic of type 2 diabetes and obesity in Western society. Infants born to diabetic women (IBDW) have alterations in cardiac morphology and function, which may predispose them to long-term adverse cardiovascular health. At present, mechanisms for adverse cardiovascular outcomes in IBDW are unknown. Abnormal maternal glucose metabolism in DM during pregnancy was previously thought to affect fetal cardiac development. However, recent findings indicate that IBDW with good 3rd trimester glucose control still develop cardiac abnormalities. In fact, other aspects of maternal nutrient metabolism and partitioning (other than glycemic control) may regulate fetal cardiac development. For example, abnormal fatty acid, triglyceride, and lipoprotein metabolism are common in DM, and maternal serum lipid levels in pregnant diabetics predict neonatal birth weight. The investigators propose that maternal fatty acid metabolism is dysregulated in diabetic pregnancy. This increases fatty acid delivery to the fetus and leads to fetal myocardial lipid accumulation, and altered neonatal heart morphology and function in IBDW. To date, this has not been explored in humans. The proposal stems from the "lipotoxicity" paradigm: chronic elevations in maternal blood lipid (i.e. fatty acid, triglyceride, very low density lipoprotein) levels during pregnancy lead to increased lipid delivery to and cause myocardial lipid deposition in the developing fetus. These lipids displace glucose utilization by the fetal myocardium; the preferred fetal heart substrate in a healthy pregnancy. Abnormal fetal heart lipid deposition and accumulation of lipid metabolic intermediates (e.g. ceramide) may lead to myocardial insulin resistance and contractile dysfunction in IBDW. The relationship between abnormal nutrient metabolism during pregnancy and adverse cardiovascular and metabolic health in diabetes may be important in other conditions such as childhood obesity in which this project could provide insight.

Specific Aims: In 25 women who have pre-gestational type 2 DM and 25 healthy non-diabetic body mass index-matched controls during the 3rd trimester of pregnancy, the investigators will address the following Aims:

Specific Aim 1: To characterize maternal lipid metabolism kinetics (fatty acid oxidation rate, lipolytic rate, fatty acid clearance rate) and maternal and fetal serum lipid concentrations (free fatty acid, triglyceride and very low density lipoprotein (VLDL)).

Hypothesis 1: Women with DM during pregnancy will have higher whole-body lipolytic rates and serum lipid concentrations, and lower whole-body fatty acid oxidation and clearance rates than healthy women without DM during pregnancy.

Specific Aim 2A: To examine the relationship among maternal lipid kinetics, maternal and fetal plasma lipid concentrations, and neonatal cardiac morphology and function in neonates born to these women.

Specific Aim 2B: To determine whether maternal lipid metabolism kinetics, maternal serum lipid levels and clinical markers of maternal glycemic control alone or in combination can predict abnormal neonatal cardiac function.

Hypothesis 2A:. Altered maternal lipid metabolism kinetics (higher lipolytic and lower fatty acid oxidation rates) will be related to elevated maternal and fetal serum lipid concentrations and abnormal neonatal cardiac function.

Hypothesis 2B. The combination of maternal lipid metabolism kinetics (lipolytic and fatty acid oxidation rates) and serum fatty acid level will be superior to markers of glycemic control (HBA1C and fructosamine) for predicting neonatal cardiac function.

Design: Whole-body lipid metabolism kinetics (fatty acid oxidation, lipolytic, clearance rates) will be measured during clinical metabolism studies using stable isotope tracer methodology and mass spectrometry performed in the Clinical Research Unit and Biomedical Mass Spectrometry Facility at Washington University School of Medicine. Umbilical cord blood will be collected at parturition and serum lipid (fatty acid, triglyceride and VLDL) and other nutrient as well as growth-related hormone levels will be quantified. Neonatal heart function (within 2 weeks of parturition) will be examined using 2D, Doppler, tissue Doppler and strain/strain rate echocardiography performed at St. Louis Children's Hospital.

Potential Impact: Currently, nothing is known regarding the role of lipid metabolism in cardiac abnormalities in IBDW. This translational proposal will address an important knowledge gap regarding the potential role of abnormal lipid metabolism in the development of cardiac abnormalities in IBDW. These associations are a critical step towards understanding the mechanisms of cardiac morphologic and functional alterations in IBDW, in order to identify clinical prognostic markers for cardiac abnormalities in IBDW, develop targeted interventions for these cardiac deficits, and to decrease the future risk of cardiovascular disease and heart failure in IBDW. The potential impact of these findings could extend not only to women and children with pre-gestational diabetes, but to other children born to women with clinical complications including gestational diabetes, obesity, intrauterine growth retardation, and HIV.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus:

  1. Women will be diagnosed with type 2 DM (pre-gestational, White classification B or C class). Since the majority of women with B or C class DM are on insulin therapy in our clinic, the investigators will recruit only women on insulin therapy (i.e. no oral diabetes medications).
  2. HbA1C ≤ 8 for greater than 3 months 32, 33.
  3. All women will have confirmed singleton pregnancies.
  4. Receive care at the Women's Health Clinic at Barnes Jewish Hospital.
  5. Pre-pregnancy BMI is anticipated to be > 30 (i.e. obese) from the data regarding the patient population of our clinic. Women with pre-pregnancy BMI between 23-40 will be included.

Control Participants:

1. No diagnosis of type 1 or 2 diabetes or previous gestational DM.
2. Women with pre-pregnancy BMI between 23-40: control participants will be BMI matched to women with DM.
3. A normal routine, standard of care 1 hour 50 gram gestational diabetes screen.
4. Receive care at the Women's Health Clinic at Barnes Jewish Hospital.
5. Patients will have a singleton pregnancy with no fetal abnormalities (as determined by routine standard of care ultrasonography).

Exclusion Criteria:

1. Multiple gestation pregnancy.
2. Oral diabetes medications.
3. Inability to provide voluntary informed consent.
4. Currently using illegal drugs (cocaine, methamphetamine, opiates).
5. Current smoker who does not agree to stop.
6. Participants with diabetes who have a BMI > 40.
7. Participants who participate in a routine (> 1x/week) exercise program.
8. History of heart disease.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants: All women who seek pre-natal care at the Women's Health Clinic Barnes Jewish Hospital in St. Louis, Missouri are screened by history at the first visit for a pre-existing diagnosis of diabetes mellitus (DM) (B or C type DM). Patients with a diagnosis of pre-gestational diabetes are transferred to a specialty clinic dedicated specifically to pre-natal care for women with diabetes. All patients with on-going pregnancies and diabetes will be approached for enrollment. Non-DM subjects have a routine screen for gestational diabetes at 24 wk gestation. After a normal result, these subjects will be approached for enrollment as controls.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2011-04; Primary Completion 2014-02 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Left ventricular strain | 1 month post partum
  Left ventricular contractility measured by speckle tracking echocardiography

SECONDARY OUTCOMES:
Maternal plasma concentration of free fatty acids during hyperinsulinemia | 3rd trimester of pregnancy
Maternal plasma interleukin-6 concentration | 3rd trimester of pregnancy
Infant birth weight | Immediately postpartum
Infant neurodevelopment | 2 years
  Bayley Scores for Infant and Toddler Motor Development
Maternal palmitate oxidation rate during hyperinsulinemia | 3rd trimester of pregnancy
  Maternal fatty acid oxidation rate measured by stable isotope tracer methodology
Maternal palmitate rate of appearance during hyperinsulinemia | 3rd trimester of pregnancy
  Maternal lipolytic rate (palmitate rate of appearance) measured by stable isotope tracer methodology

CONTACTS AND LOCATIONS:
Overall Officials: William T Cade, PT, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Result] Cade WT, Tinius RA, Reeds DN, Patterson BW, Cahill AG. Maternal Glucose and Fatty Acid Kinetics and Infant Birth Weight in Obese Women With Type 2 Diabetes. Diabetes. 2016 Apr;65(4):893-901. doi: 10.2337/db15-1061. Epub 2016 Feb 9. PMID 26861786